CLINICAL TRIAL: NCT03184272
Title: Accuracy of Non-invasive Assessment of Cardiac Output and Fluid Responsiveness in Patients Undergoing Bariatric Procedures.
Brief Title: Non-invasive Assessment of Cardiac Output and Fluid Responsiveness in Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Dr. Jochen Renner, Clinical Professor, University Hospital Schleswig-Holstein
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IN-BAR-01
Record Dates: First submitted 2017-06-03; First posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Bariatric Surgery; Hemodynamics
Keywords: limitation in conventional monitoring
MeSH Terms: interventions — Equipment and Supplies; BaseLine dental cement

STUDY DESIGN:
Intervention Model Description: evaluate direct impacts of preventive measurement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bariatric surgery (Experimental): baseline alert 1; Anti-Trendelenburg-position (ATB); Anti-Trendelenburg-position (ATB) in narcosis; baseline in narcosis 1; passive leg raising; volume bolus substitution (15 ml/kgKG Sterofundin balanced solution); baseline in narcosis 2; start capnoperitoneum; Anti-Trendelenburg-position (ATB) plus capnoperitoneum; ATB plus capnoperitoneum plus volume bolus substitution (15 ml/kgKG Sterofundin balanced solution); ATB loss of capnoperitoneum; baseline in narcosis; baseline alert 2; torso position rising 30° at the beginning; torso position rising 30° at the end
  Interventions: Procedure: baseline alert 1; Procedure: Anti-Trendelenburg-position (ATB); Procedure: ATB in narcosis; Procedure: baseline in narcosis 1; Procedure: passive leg raising; Procedure: volume bolus substitution; Procedure: baseline in narcosis 2; Procedure: start capnoperitoneum; Procedure: ATB plus capnoperitoneum; Procedure: ATB plus capnoperitoneum plus volume bolus substitution; Procedure: ATB loss of capnoperitoneum; Procedure: baseline; Procedure: baseline alert 2; Procedure: torso position rising 30° at the beginning; Procedure: torso position rising 30° at the end

INTERVENTIONS:
Procedure: baseline alert 1 — measurement in supine position
  Other Names: Device; Nexfin© vs FloTrac© vs sphygmomanometric blood pressure
Procedure: Anti-Trendelenburg-position (ATB) — measurement under ATB
  Other Names: Device; Nexfin© vs FloTrac© vs sphygmomanometric blood pressure
Procedure: ATB in narcosis — measurement under ATB in narcosis
  Other Names: Device; Nexfin© vs FloTrac© vs sphygmomanometric blood pressure
Procedure: baseline in narcosis 1 — measurement in supine position in narcosis
  Other Names: Device; Nexfin© vs FloTrac© vs sphygmomanometric blood pressure
Procedure: passive leg raising — measurement under passive leg raising
  Other Names: Device; Nexfin© vs FloTrac© vs sphygmomanometric blood pressure
Procedure: volume bolus substitution — measurement in supine position after volume bolus (15 ml/kgKG Sterofundin balanced solution intravenous)
  Other Names: Device
Procedure: baseline in narcosis 2 — measurement in supine position
  Other Names: Nexfin© vs FloTrac© vs sphygmomanometric blood pressure
Procedure: start capnoperitoneum — measurement in supine position
  Other Names: Device; Nexfin© vs FloTrac© vs sphygmomanometric blood pressure
Procedure: ATB plus capnoperitoneum — measurement under ATB plus capnoperitoneum
  Other Names: Device; Nexfin© vs FloTrac© vs sphygmomanometric blood pressure
Procedure: ATB plus capnoperitoneum plus volume bolus substitution — measurement in ATB plus capnoperitoneum after volume bolus (15 ml/kgKG Sterofundin balanced solution intravenous)
  Other Names: Device; Nexfin© vs FloTrac© vs sphygmomanometric blood pressure
Procedure: ATB loss of capnoperitoneum — measurement under ATB
  Other Names: Device; Nexfin© vs FloTrac© vs sphygmomanometric blood pressure
Procedure: baseline — measurement in supine position
  Other Names: Device; Nexfin© vs FloTrac© vs sphygmomanometric blood pressure
Procedure: baseline alert 2 — measurement in supine position
  Other Names: Device; Nexfin© vs FloTrac© vs sphygmomanometric blood pressure
Procedure: torso position rising 30° at the beginning — measurement in the recovery unit
  Other Names: Device; Nexfin© vs FloTrac© vs sphygmomanometric blood pressure
Procedure: torso position rising 30° at the end — measurement in the recovery unit
  Other Names: Device; Nexfin© vs FloTrac© vs sphygmomanometric blood pressure

SUMMARY:
Comparability of discontinuous non-invasive (sphygomanometric) and continuous semi-invasive and invasive (Masimo©; Nexfin© Monitoring ; FloTrac © Edwards Lifesciences) beat to beat measurement methods for the determination of cardiac output and fluid responsiveness in patients undergoing bariatric surgery.

DETAILED DESCRIPTION:
Comparability of discontinuous non-invasive (sphygomanometric) and continuous semi-invasive and invasive (Masimo©; Nexfin© Monitoring ; FloTrac © Edwards Lifesciences) beat to beat measurement methods for the determination of cardiac output and fluid responsiveness in patients undergoing bariatric surgery.

Bariatric patients show limitations regarding the conventional monitoring options with ECG derivation, pulse oxymetric oxygen saturation and sphygmo-manometric blood pressure measurement. From a clinical point of view this results in an invasive arterial blood pressure monitoring. In addition to that, intraoperative extreme changes of the patients position on the table combined with the applied pneumoperitoneum during the minimally invasive laparoscopic surgery can significantly influence the cardiovascular parameters. An invasive arterial blood pressure monitoring is able to reproduce the blood pressure by stroke, but it does not give any information about the cardiac output. The sphygmomanometric blood pressure measurement also entails the risk of insufficient detection of a hypotonic phase in the measurement. Additional monitoring systems are currently available, which are capable of measuring completely non-invasive or semi-invasively different cardiovascular parameters such as cardiac output (CO) and volume responsiveness. In this study, the investigators will compare continuous and discontinuous cardiovascular monitoring procedures and their parameters. The measurements take place at specific times, under defined changes in the body position with the additional influence of the pneumoperitoneum.

These changes are recorded and compared at the same time during different measuring methods preoperatively, intraoperatively and postoperatively. The non-invasive Nexfin © Monitoring (Edwards Lifesciences) is to be evaluated and compared with further measurement methods (FloTrac © (Edwards Lifesciences)) as well as the sphygmomanometric upper arm blood pressure measurement. The investigators also compare the non-invasive and invasive continuous beat to beat blood pressure measurement with conventional, discontinuous sphygomanometric upper arm blood pressure measurement.

The planned study is the comparison of 3 different hemodynamic monitoring procedures. For the evaluation we use the method used by Bland and Altmann for calculating the mean deviation (bias) and the precision (mean value ± 2 standard deviations. In the case of multiple measurements , the modification of the Bland-Altman method is applied (repeated measurements). The number of cases was determined with n = 60 patients, followed by an intermediate evaluation. For a Bland-Altman analysis, the width w of the confidence interval for the Limits of Agreement is calculated as w = 6.79 • σ • 1 / √n, where n is number of cases and σ is the standard deviation. For a case count of n = 60, the result is w = 0.88 • σ and thus for this explorative study a sufficiently large number. In case of the dynamic variables, the percentage matching and the calculation of the kappa index are also used for the statistical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Indication for bariatric surgery was made
* Classification according to the American Society of Anesthesiologists (ASA) 2-4
* Age > 18 years
* Elective laparoscopic surgery
* Written declaration of consent
* Body Mass Index > 30 kg / m²

Exclusion Criteria:

* atrial fibrillation
* cardiac arrhythmias
* aortic aneurysm > 4,5 cm
* Peripheral arterial occlusive desease grade 3-4
* age < 18 years
* missing or incorrect patient consent form
* cognitive or linguistic barriers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Non-invasive cardiac output, i.e. stroke volume measurement using Nexfin technology | From the beginning of surgery to admission to the PACU, approximately 4 hours
  Accuracy of non-invasive assessment of cardiac output, i.e. stroke volume index in comparison to an invasive standard using FloTrac Vigileo technology

SECONDARY OUTCOMES:
Non-invasive assessment of fluid responsiveness using Nexfin technology | From the beginning of surgery to admission to the PACU, approximately 4 hours
  Accuracy of non-invasive assessment of fluid responsiveness (PPV, SVV) in comparison to an invasive standard using FloTrac Vigileo technology

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Schleswig-Holstein Campus Kiel - Klinik für Anästhesiologie und Operative Intensivmedizin, Kiel, Deutschland (deu), Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lorenzen U, Pohlmann M, Hansen J, Klose P, Gruenewald M, Renner J, Elke G. Perioperative non-invasive versus semi-invasive cardiac index monitoring in patients with bariatric surgery - a prospective observational study. BMC Anesthesiol. 2020 Aug 10;20(1):196. doi: 10.1186/s12871-020-01110-x. PMID 32778047